CLINICAL TRIAL: NCT01857466
Title: Additional Benefit of Hemostatic Sealant in Preserving Ovarian Reserve During Laparoscopic Ovarian Cystectomy: a Randomized Controlled Trial
Brief Title: Ovarian Reserve After Ovarian Hemostasis by Floseal Matrix
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: CHA University (Other)
Responsible Party: Principal Investigator, Taejong Song, Professor, CHA University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KNC13-017
Record Dates: First submitted 2013-05-16; First posted 2013-05-20 (Estimated); Last update posted 2014-06-25 (Estimated); Status verified 2014-06

CONDITIONS: Ovarian Cysts
MeSH Terms: conditions — Ovarian Cysts | interventions — FloSeal Matrix

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Floseal (Experimental): In the Floseal group, the sites of bleeding were covered with Floseal under direct vision with a laparoscopic applicator and ovarian cortex was closed on itself and waited for 2 minutes for Floseal to act. Then, subsequently bleeding sites were reexamined with irrigation.
  Interventions: Procedure: Floseal
- Bipolar coagulation (Active Comparator): In the bipolar group, hemostasis of the ovarian parenchyma was achieved with selective minimal (20-30 watt current) bipolar coagulation without excessive coagulation of surgical defect to avoid damaging the ovary.
  Interventions: Procedure: Bipolar coagulation

INTERVENTIONS:
Procedure: Floseal
  Arms: Floseal
Procedure: Bipolar coagulation
  Arms: Bipolar coagulation

SUMMARY:
Laparoscopy has become the gold standard for the surgical treatment of benign ovarian cysts and is usually performed by stripping the ovarian cyst wall, followed by bleeding control of the ovarian wound ground using bipolar coagulation. However, the hemostasis with bipolar coagulation could result in the damage of ovarian reserve and decrease the response of the ovaries to hormonal stimulation for assisted reproductive technologies. The possible mechanism may contribute to thermal destruction of ovarian follicles by excessive use of bipolar coagulation for hemostasis purposes.

To avoid additional ovarian tissue damage by conventional bipolar coagulation being potentially important ovarian reproductive function, hemostasis using various topical hemostatic agents has introduced to control post-cystectomy ovarian wound bleeding. Among them, FloSeal (Baxter Healthcare Corporation, Deerfield, IL, USA) is a hemostatic matrix sealant composed of a gelatin-based matrix and thrombin solution. On coming into contact with blood after application at a bleeding site, the gelatin particles swell and tamponade bleeding. The bulk of the gelatin matrix-thrombin composite has the effect of slowing blood flow and providing exposure to a high thrombin concentration, thus hastening clot formation. Therefore, it may more suitable for use in post-cystectomy ovarian wound bleeding, where there is superficially pervasive focus of bleeding.

Ovarian reserve is defined as the functional potential of the ovary, which reflects the number and quality of antral follicles left in the ovary, and is correlated with the response to ovarian stimulation using exogenous gonadotropin. Serum anti-Müllerian hormone (AMH) has been accepted as the most reliable and easily measurable marker for postoperative assessment of ovarian reserve.

The investigators conducted a multicenter, large-scale, randomized controlled trial to investigate whether hemostasis by Floseal was superior to that by bipolar coagulation in preserving ovarian reserve by assessing serial AMH levels in patients undergoing laparoscopic ovarian cystectomy for benign ovarian cysts.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 45 years
* maximum diameter of the cyst between 3 and 10 cm
* regular menstrual bleeding (defined as cycle length less than 21 or more than 45 days)
* appropriate medical status for laparoscopic surgery (American Society of Anesthesiologists Physical Status classification 1 or 2).

Exclusion Criteria:

* any suspicious finding of malignant ovarian diseases
* postmenopausal status
* baseline serum AMH < 0.50 ng/mL
* pregnancy
* lactation
* any other endocrine diseases (such as thyroid dysfunction, hyperprolactinemia, or Cushing's syndrome)
* use of hormonal treatments in the 3 months before enrollment

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2012-12; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Decline rate of serum AMH levels | 3 months after therapy
  The primary outcome of the study was the impact on ovarian reserve determined by serum AMH levels after the applications of two hemostatic techniques for ovarian wound bleeding.

CONTACTS AND LOCATIONS:
Overall Officials: Taejong Song, M.D, Principal Investigator — CHA Gangnam Medical Center, Seoul, Republic of Korea
Locations (3):
- South Korea (3):
  - National Health Insurance Service Ilsan Hospital, Goyang
  - CHA Gangnam Medical Center, Seoul
  - Kangbuk Samsung Hospital, Sungkyunkwan University, Seoul

REFERENCES:
- [Derived] Song T, Lee SH, Kim WY. Additional benefit of hemostatic sealant in preservation of ovarian reserve during laparoscopic ovarian cystectomy: a multi-center, randomized controlled trial. Hum Reprod. 2014 Aug;29(8):1659-65. doi: 10.1093/humrep/deu125. Epub 2014 Jun 4. PMID 24903197